CLINICAL TRIAL: NCT05075291
Title: Repeated Suicide Attempts in a Patient Suffering From Addiction to Tramadol: a Case Report
Brief Title: Suicide Attempts and Tramadol : a Case Report
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0571
Record Dates: First submitted 2021-09-18; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Suicide, Attempted; Addiction
Keywords: Suicide; Addiction; Opioids
MeSH Terms: conditions — Suicide, Attempted; Behavior, Addictive; Suicide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, over the last years the use weak opioid analgesics decreased́, whereas that of strong opioid analgesics (OFMA). Hospitalizations for opioid overdose increased́ by 128% from 2000 to 2015, and deaths related to prescribed opioid overdose increased significantly, by 161%, from 2000 to 2014.In addition, recent studies suggest a link between opioid system dysfunction and suicidal behavior.

In parallel, studies are emerging showing the potential interest of using Tramadol as an antidepressant. Indeed, this opiate analgesic also acts on the serotonergic and dopaminergic systems, and would have an antidepressant effect.Thus, the investigators can legitimately wonder whether the use of Tramadol as an antidepressant might not pose a problem in patients at risk of suicide.

This study aims to describe a clinical case of a patient hospitalized in the Department of Psychiatric Emergency and Post-Emergency (Montpellier University Hospital) who developed a severe addiction to Tramadol (consumption up to 5 times the maximum recommended dose per day) and evaluate whether this may have increased her suicidal risk, in order to warn prescribers about the suicidal risk of Tramadol.

ELIGIBILITY:
Inclusion criteria:

* Multiple suicide attempts
* Tramadol addiction

NA : patient case report

Exclusion criteria:

- None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A single patient with multiple suicide attempts related to her addiction to Tramadol.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Lifetime suicidal events | day 1
  Occurrence of suicidal events (actuel, interrupted and aborted or self-aborted suicide attempts) based on the patient medical records.

SECONDARY OUTCOMES:
Depressive symptomatology | day 1
  Depressive symptomatology assessed with the Montgomery Asberg Depression Rating Scale (MADRS). The total score ranges from 0 to 60 :
  * scores between 0 and 6 : no depression,
  * scores between 7 and 19 : mild depression,
  * scores between 20 and 34 : moderate depression
  * scores above 34 : severe depression
Suicidal ideation | day 1
  Suicidal thoughts assessed with the Columbia Suicide Severity Scale (C-SSRS). The suicidal ideation severity subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each one ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Psychological pain | day 1
  Psychological pain assessed with a Likert scale : Strongly disagree, Disagree, Neutral, Agree, Strongly agree
Anxiety | day 1
  Anxiety level assessed with a Likert scale : Strongly disagree, Disagree, Neutral, Agree, Strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte NOBILE, PharmD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC